CLINICAL TRIAL: NCT00974337
Title: Basal and Stimulated Cortisol Levels in Preterm Very Low Birth Weight Infants With and Without Shock: A Cross-sectional Study
Brief Title: Relative Adrenal Insufficiency in Preterm Very Low Birth Weight Infants With Shock
Status: Completed | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, M. Jeeva Sankar, Assistant Professor, All India Institute of Medical Sciences
Other Study IDs: A-123/2008
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal insufficiency; cortisol; preterm; shock; neonate
MeSH Terms: conditions — Adrenal Insufficiency; Premature Birth; Shock

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shock: Preterm VLBW infants with shock (BP <3rd centile for gestation and birth weight with at least one of the following:
  1. Prolonged capillary refill time (>3sec)
  2. Reduced urine output (<1 mL/kg/hr)
  3. Metabolic acidosis (Base deficit >5)
- No shock: Hemodynamically stable infant with normal blood pressure, capillary refill time, and urine output

SUMMARY:
The objective of this study is to estimate the prevalence of relative adrenal insufficiency in preterm very low birth weight infants with and without shock.

DETAILED DESCRIPTION:
Till date, no studies are available that have evaluated the incidence of relative adrenal insufficiency in preterm very low birth weight (VLBW) infants with shock. The focus had been on stable preterm and critically ill preterm infants. Given that steroid treatment improves blood pressure and stabilizes cardiovascular status in preterm infants with volume and pressor-resistant hypotension,it becomes essential to examine the incidence of adrenal insufficiency in this cohort (rather than a broad group of critically ill preterm infants). Moreover, there are no studies on adrenal function in Indian neonates.

The purpose of this study is to compare the levels of basal and stimulated (using low dose [1µg/k] ACTH) cortisol levels in preterm (28-34 weeks gestation) very low birth weight (birth weight 750 gm to 1500 gm) infants with shock in the first week of life requiring vasopressor therapy and matched (gestation, birth weight, postnatal age-matched) hemodynamically stable infants ('control group').

ELIGIBILITY:
Inclusion Criteria:

* All preterm (28 to 34 week gestation) very low birth weight (birth weight 750-1500grams.) infants born at AIIMS would be eligible for enrollment in the study. Of these infants, those who meet the following criteria would be enrolled.
* Cases: Preterm (28 to 34 week gestation) infants with birth weight between 750 and 1500 grams with shock in the first week of life requiring vasopressor therapy (dopamine or dobutamine or both in a dose of > 10 mcg/kg/min)
* Controls: Stable preterm (28 to 34 week gestation) infants with birth weight between 750 and 1500 grams who are matched for gestational age, birth weight, postnatal-age.

Exclusion Criteria:

* Major congenital malformations
* Mother receiving anticonvulsant / anti-tubercular drugs (rifampicin, isoniazid)
* Postnatal corticosteroid treatment
* Refusal to give consent

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm (28 to 34 week gestation) very low birth weight (birth weight 750-1500grams) infants born at AIIMS
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Baseline cortisol | At enrollment
Stimulated cortisol (after ACTH stimulation) | 30 minutes after ACTH stimulation

SECONDARY OUTCOMES:
Survival till discharge or day 28 of life | Until discharge or 28 days of life
Chronic lung disease (CLD) | 36 weeks postmenstrual age
Sepsis | until 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Paul, MD PhD, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Suman Sarkar, MBBS, Principal Investigator — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Mari J Sankar, MD DM, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Ramesh Agarwal, MD DM, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India